CLINICAL TRIAL: NCT01327950
Title: EPIC SFA - Physician Initiated Trial Investigating the Efficacy of the EPICTM Nitinol Vascular Stent System (Boston Scientific) in Superficial Femoral Lesions: A Prospective, Multi-center Non- Randomized Study - Endoconsul 003
Brief Title: Efficacy of the EPIC Nitinol Vascular Stent System in Superficial Femoral Artery (SFA) Lesions
Acronym: EPIC SFA BR
Status: Completed | Type: Observational
Sponsor: Endovascular Consultoria Limitada (Industry)
Collaborators: Boston Scientific Corporation (Industry); Angiolog Consultoria Ltda (Unknown)
Responsible Party: Sponsor
Other Study IDs: EPIC SFA Brazil - ISROTH10003
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Superficial Femoral Artery Stenosis; Atherosclerosis of Femoral Artery
Keywords: Percutaneous treatment; Superficial Femoral Artery lesions; EPIC Nitinol Vascular Stent System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Superficial Femoral Lesions: Patients undergoing percutaneous treatment of Superficial Femoral Artery lesions

SUMMARY:
This is a national, prospective, multi-center, non-randomized study to evaluate the long-term efficacy and integrity of the EPICTM Nitinol Vascular Stent System in Superficial Femoral Artery (SFA) lesions. A total of 100 patients will be included in approximately 10 sites. The study is designed to demonstrate the EPIC Nitinol Vascular Stent System is non- inferior to the published patency rates found in the literature. This non-inferiority will be established by proving that the true rate for the EPICTM Nitinol Vascular Stent System is higher than 82% minus a 10% delta.

ELIGIBILITY:
General Inclusion Criteria:

* Patient presenting with a stenosis, re-stenosis after PTA (or adjunct therapy, excluding stents or stent grafts) or occlusion in the native superficial femoral artery (SFA), or SFA and proximal popliteal artery, suitable for primary stenting;
* Patient has a score from 2 to 5 following Rutherford classification;
* Patient is willing to comply with specified follow-up evaluations at the specified times;
* Patient is at least 18 years old; - Patient (or their legal representative) understands the nature of the procedure and provides written informed consent prior to enrollment in the study;
* Patient is eligible for treatment with the self-expanding EPIC Nitinol Vascular Stent System

Notes:

* If the patient has a contralateral peripheral lesion,this lesion can be treated as a non-target lesion before or after the study procedure
* If the patient has an ipsilateral iliac lesion,the lesion can be treated as a non target lesion, if the treatment is conducted before the target lesion treatment (during the same procedure or during a previous procedure), with a successful result defined as less than 30% residual diameter stenosis

Angiographic Inclusion Criteria:

* Target lesion(s) location is situated in the native SFA or SFA and proximal popliteal artery, with its most proximal point at least 1cm below the origin of the deep femoral artery and its distal point at least 3cm proximal to the knee joint, as measured by ipsilateral oblique view for proximal lesions and straight posterioanterior (PA) view for distal lesions;
* Evidence of at least 50% stenosis, re-stenosis after PTA (or adjunct therapy, excluding stents or stent grafts) or occlusion in the target lesion;
* Target lesion(s) total length is minimally 4cm and maximally 11cm and is amenable to treatment with a single stent;
* Target vessel diameter visually estimated is > 4mm and < 6.5mm
* There is angiographic evidence of at least one-vessel-runoff to the foot

General Exclusion Criteria:

* Presence of another stent or stent graft in the target vessel that was placed during a previous procedure;
* Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis;
* Previous bypass surgery in the same limb; - Necessity to treat target vessel with more than one EPICTM stent;
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated;
* Patient has bleeding diathesis, coagulopathy, known hypercoagulable condition or refuses blood transfusion;
* Patients with known hypersensitivity to nickel-titanium;
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding;
* Life expectancy of less than twelve months;
* Ipsilateral iliac treatment before the target lesion procedure with a residual stenosis > 30% or ipsilateral iliac treatment conducted after the target lesion procedure;
* Use of cutting balloon, scoring balloon, thrombectomy, arthrectomy, brachytherapy or laser devices during procedure;
* Any patient considered to be hemodynamically unstable at onset of procedure;
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period;
* Patient presenting one of the following comorbid conditions: hemodialysis, elevated creatine levels (> 2.5mg/dl), recent MI or hemorrhagic stroke occurrence (both within 30 days).

Angiographic Exclusion Criteria:

* Inability to cross the target lesion by means of an exchangeable guidewire and to re-enter the true vessel lumen distal to the lesion site;
* Presence of a significant (minimally 50%) stenosis or occlusion in the ipsilateral common femoral artery;
* Aneurysm located at the level of the to-be-treated artery; - Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site; - Perforation (evidenced by extravasation of contrast medium), dissection or other injury of the access or target vessel requiring additional stenting or surgery prior to the start of the index procedure;
* Focal popliteal artery disease in the absence of femoral disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing percutaneous treatment of Superficial Femoral Artery lesions
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the long-term efficacy and integrity of the EPICTM Nitinol Vascular Stent System in SFA lesions. | 12 months
  The primary endpoint is primary patency rate at 12 months as determined by Duplex ultrasound at twelve months, defined as a target vessel with <50% diameter stenosis at twelve months (systolic velocity ratio no greater than 2.4), without occurrence of target lesion revascularization between the index procedure and the twelve months follow-up control

SECONDARY OUTCOMES:
Initial arteriographic success | immediately following stent implantation (day 1)
  Initial arteriographic success, defined as arteriographic evidence of improvement in luminal diameter to <30% residual stenosis and/or an increase of at least 50% in luminal diameter immediately following stent implantation;
Primary patency rate | 6 months
  Primary patency rate at 6 months as determined by Duplex ultrasound at six months, defined as a target vessel with <50% diameter stenosis at six months (systolic velocity ratio no greater than 2.4), without occurrence of target lesion revascularization between the index procedure and the twelve months follow-up control;
Major adverse event | 1 year
  - Major adverse event rate at 1 year, defined as: clinically- driven TLR, major amputation, all-cause mortality;
Technical Success | immediately following stent implantation (day 1)
  - Technical success, defined as the ability to cross the target lesion with the device and deploy the stent as intended at the treatment site;
Increase of ABI | 1 year
  - Increase of Ankle-Brachial Index (ABI) at 1 year, defined as: an increase in ABI compared to baseline.

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Instituto de Medicina Integral Professor Fernando Figueira (IMIP), Recife, Pernambuco
  - Clinica Coris Medicina Avançada /Baia Sul Medical Center, Florianópolis, Santa Catarina
  - Hospital Santa Marcelina de São Paulo, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Irmandade Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo